CLINICAL TRIAL: NCT03687255
Title: A Phase 3, Randomized, Double-Blind, Study to Evaluate the Efficacy and Safety of Cefepime-AAI101 Compared to Piperacillin/Tazobactam in the Treatment of Complicated Urinary Tract Infections, Including Acute Pyelonephritis.
Brief Title: Safety and Efficacy Study of Cefepime-AAI101 in the Treatment of Complicated Urinary Tract Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allecra (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-301
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cefepime; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cefepime/AAI101 combination (Experimental): Cefepime 2 g in combination with AAI101 500 mg q8h (2 hour infusion)
  Interventions: Drug: cefepime/AAI101 combination
- piperacillin/tazobactam (Active Comparator): Piperacillin 4 g in combination with Tazobactan 500 mg q8h (2 hour infusion)
  Interventions: Drug: Piperacillin/tazobactam

INTERVENTIONS:
Drug: cefepime/AAI101 combination — cefepime 2 g / AAI101 500 mg
  Arms: cefepime/AAI101 combination
Drug: Piperacillin/tazobactam — piperacillin 4 GM / tazobactam 500 MG
  Other Names: PIP/TAZ
  Arms: piperacillin/tazobactam

SUMMARY:
Multi-center, randomized, double-blind, non-inferiority study of cefepime 2 g/AAI101 500 mg combination compared to piperacillin 4 g/tazobactam 500 mg in a population of adult patients with cUTI or AP. The study will be conducted in approximately 115 sites located in the EU, the US, Central, South America and South Africa.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients >18 years of age at the time of signing of informed consent;
2. Expectation that the patient's cUTI or AP will require hospitalisation and initial treatment with at least 7 days of intravenous (i.v.) antibiotics;
3. Female patients who are no longer of childbearing potential
4. Female patients of childbearing potential must have a negative urine and/or serum pregnancy test (serum β-human chorionic gonadotropin) within 1 day prior to study entry;
5. Male patients, female patients receiving hormone replacement therapy (HRT), and female patients of childbearing potential must agree to use highly effective contraception methods
6. Pyuria, defined as: a. White blood cell count >10 cells/mm3 in unspun urine or ≥10 cells/high power field in spun urine sediment; or b. Urinalysis/dipstick analysis positive for leukocyte esterase;
7. Clinical signs and/or symptoms of cUTI or AP
8. Have a baseline urine culture specimen obtained within 48 hours prior to randomization
9. Expectation, in the judgment of the Investigator, that any implanted urinary instrumentation (e.g., nephrostomy tubes, ureteric stents, etc.) will be surgically removed or replaced before or within 24 hours after randomisation, unless removal or replacement is considered unsafe or contraindicated.

Exclusion Criteria

1. Known urine culture with Gram-positive primary pathogen at ≥105 colony-forming units (CFU)/mL (not contaminant) or suspected Gram-positive pathogen by Gram staining (Note: Gram staining is optional);
2. History of significant hypersensitivity or allergic reaction to cefepime, piperacillin/tazobactam, any of the excipients used in the respective formulations, any beta-lactam antibiotics (e.g., cephalosporins, penicillins, carbapenems, or monobactams), or any beta-lactamase inhibitors (e.g., tazobactam, sulbactam, or clavulanic acid);
3. In the opinion of the Investigator, the patient is considered unlikely to survive the approximately 6-week study period;
4. Weight >180 kg;
5. Concurrent infection that would interfere with evaluation of response to the study antibiotics;
6. Need for or receipt of concomitant systemic antimicrobial agents after signing of informed consent, in addition to those designated in the study-treatment groups, with the exception of a single oral dose of any antifungal treatment for vaginal candidiasis;
7. Receipt of potentially effective systemic antibacterial therapy for a continuous duration of > 24 hours during the previous 72 hours before the study-qualifying baseline urine is obtained;
8. Complicated urinary tract infection (UTI) known at study entry to be caused by pathogens resistant to the study antibiotics;
9. Likely to require the use of an antibiotic for cUTI or AP prophylaxis during the patient's participation in the study;
10. Intractable UTI at baseline that the Investigator anticipates would require >14 days of study drug therapy;
11. Complete, permanent obstruction of the urinary tract that is not anticipated to be medically or surgically relieved during i.v. study therapy and before End of Treatment (EOT);
12. Gross hematuria requiring intervention other than administration of study drug or removal or exchange of a urinary catheter;
13. Presence of any known or suspected disease or condition that, in the opinion of the Investigator, may confound the assessment of efficacy.
14. Suspected or confirmed acute bacterial prostatitis, orchitis, epididymitis, or chronic bacterial prostatitis as determined by history and/or physical examination;
15. Impairment of renal function with estimated glomerular filtration rate <30 mL/min/1.73 m2 calculated by the 4-variable Modification of Diet in Renal Disease study equation,
16. Urinary tract surgery within 7 days prior to randomisation or urinary tract surgery planned during the study period (except surgery required to relieve an obstruction or place a stent or nephrostomy prior to EOT);
17. Any condition or circumstance that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of study data;
18. Any rapidly progressing disease or immediately life-threatening illness, including acute hepatic failure and respiratory failure;
19. Presence of sepsis, producing life-threatening organ dysfunction
20. A QT interval corrected using Fridericia's formula >450 msec;
21. Immunocompromising condition, including known history of acquired immune deficiency syndrome or known recent CD4 count <200/mm3, hematological malignancy, or bone marrow transplantation; or immunosuppressive therapy including cancer chemotherapy, medications for prevention of organ transplantation rejection, or the administration of corticosteroids ≥20 mg of prednisone or equivalent per day administered continuously for >14 days prior to randomisation;
22. One or more of the following laboratory abnormalities in baseline specimens obtained at Screening: aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or total bilirubin level >3 × upper limit of normal, or current clinically significant liver disease, including any form of known liver cirrhosis;
23. One or more of the following laboratory abnormalities at Screening: platelet count <50,000/μL, absolute neutrophil count <1,000/mm3, or hemoglobin <8 g/dL;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1043 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in the Microbiological Modified Intent to Treat (m-MITT) Population who achieve overall treatment success at Test Of Cure (TOC) | 7 days after EOT [±2 days] for patients receiving 7 days of treatment and 19 days after randomization [±2 days] for patients receiving more than 7 days of treatment.
  Treatment success is defined as the composite of clinical outcome of Cure and the microbiological outcome of Eradication (<103 CFU/mL in urine culture).

SECONDARY OUTCOMES:
Proportion of patients in the m-MITT Population with overall treatment success at End of Treatment (EOT) | 7 days for patients with cUTI only and up to 14 days for patients cUTI and blood stream infections
  Treatment success is defined as the composite of clinical outcome of Cure and the microbiological outcome of Eradication (<103 CFU/mL in urine culture).

CONTACTS AND LOCATIONS:
Locations (24):
- United States (6):
  - St. Josephs Clinical Research, Anaheim, California
  - Southbay Pharma Research, Buena Park, California
  - Florida Urology Partners, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
- HIGA Dr Ramon Carrillo, Buenos Aires, Argentina
- Brest Regional Hospital, Brest, Belarus
- MHAT Rahila Angelova AD, Pernik, Pernik, Bulgaria
- University Hospital for Infectious Diseases "Dr. Fran Mihaljevic" Department for general infectious diseases, Zagreb, Croatia
- Tartu University Hospital, Tartu, Estonia
- Unimed Adjara - Kutaisi oncological centre, Kutaisi, Georgia
- Bugat Pal Korhaz, Gyöngyös, Hungary
- Uroklinika, LLC, Riga, Latvia
- Republican Siauliai caunty hospital, Šiauliai, Lithuania
- Centro Especializado en Investigación Clínica S.C., Boca del Río, Mexico
- Clinica Internacional - Sede San Borja, Lima, Peru
- Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Klinika Chorob Wewnetrznych, Nefrologii i Transplantologii, Warsaw, Poland
- Scientific Research Center Eco-Safety, Saint Petersburg, Russia
- Clinical Hospital Center Zvezdara, Belgrade, Serbia
- Interne oddelenie, Nemocnica Malacky, Nemocnicna a.s., Malacky, Slovakia
- Clinical Projects Research, Worcester, South Africa
- Hospital del Mar, Department of Infectious Disease, Barcelona, Spain
- Chernihiv City Hospital #2 of Chernihiv City Council, department of Urology, Chernihiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaye KS, Belley A, Barth P, Lahlou O, Knechtle P, Motta P, Velicitat P. Effect of Cefepime/Enmetazobactam vs Piperacillin/Tazobactam on Clinical Cure and Microbiological Eradication in Patients With Complicated Urinary Tract Infection or Acute Pyelonephritis: A Randomized Clinical Trial. JAMA. 2022 Oct 4;328(13):1304-1314. doi: 10.1001/jama.2022.17034. PMID 36194218